CLINICAL TRIAL: NCT07188038
Title: The Impact of Low Versus High Positive End-Expiratory Pressure on Diaphragm Function, Ventilation Efficiency, and Lung Mechanics During Pressure Support Ventilation: A Randomized Interventional Crossover Study
Brief Title: The Impact of Low Versus High Positive End-expiratory Pressure on Diaphragm Function, Ventilation Efficiency, and Lung Mechanics
Acronym: INFLATE-ICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Sahlgrenska University Hospital (Other); Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-01286-01
Record Dates: First submitted 2025-09-01; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Failure; ARDS (Acute Respiratory Distress Syndrome); Pneumonia; Respiratory Insufficiency
Keywords: Positive end-expiratory pressure; PEEP; pressure support ventilation; assisted breathing; Inspiratory effort; Inspiratory drive; Ventilation efficiency; Diaphragm
MeSH Terms: conditions — Respiratory Insufficiency; Acute Lung Injury; Pneumonia

STUDY DESIGN:
Intervention Model Description: Randomized interventional crossover study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low PEEP (Experimental): Low positive end-expiratory pressure (4 cmH2O)
  Interventions: Procedure: Low positive end-expiratory pressure
- Medium PEEP (Experimental): Medium positive end-expiratory pressure (10 cmH2O)
  Interventions: Procedure: Medium positive end-expiratory pressure
- High PEEP (Experimental): High positive end-expiratory pressure (16 cmH2O)
  Interventions: Procedure: High positive end-expiratory pressure

INTERVENTIONS:
Procedure: Low positive end-expiratory pressure — Low (4 cmH2O) positive end-expiratory pressure (PEEP) will be applied during pressure support ventilation. The PEEP level will be kept for 10 minutes prior to data acquisition.
  Arms: Low PEEP
Procedure: Medium positive end-expiratory pressure — Medium (10 cmH2O) positive end-expiratory pressure (PEEP) will be applied during pressure support ventilation. The PEEP level will be kept for 10 minutes prior to data acquisition.
  Arms: Medium PEEP
Procedure: High positive end-expiratory pressure — High(16 cmH2O) positive end-expiratory pressure (PEEP) will be applied during pressure support ventilation. The PEEP level will be kept for 10 minutes prior to data acquisition.
  Arms: High PEEP

SUMMARY:
The goal of this interventional study is to evaluate the effect of different positive end-expiratory pressures (PEEP) on lung and diaphragm function in patients mechanically ventilated with pressure support ventilation in the intensive care unit. The main questions aim to answer:

Does higher PEEP level affect diaphragm contractions and ventilatory efficiency? Does higher PEEP level limit inspiratory efforts? Does higher PEEP level affect lung compliance?

The participants will be subjected to three different PEEP levels during pressure support ventilation:

Low PEEP (4 cmH2O), Medium PEEP (10 cmH2O), High PEEP (16 cmH2O).

The lung and diaphragm function will be evaluated using high-resolution esophageal manometry, electrical activity of the diaphragm, external diaphragm ultrasound and spirometric ventilator data.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation with pressure support or mechanical ventilation with possibility to transition to pressure support
* Oxygen requirement ≤ 50%
* Pressure support ≤ 12 cmH2O
* PEEP ≤ 12 cmH2O
* Age ≥ 18 years
* Adequate intravascular volume status

Exclusion Criteria:

* Circulatory instability
* Brain death diagnosis/brain death evaluation
* Norepinephrine dose > 0.4 µg/kg/min
* Muscle relaxation administered within 2 hours
* Pregnancy
* Contraindication to esophageal catheterization (e.g., esophageal varices)
* Conditions with increased risk of pneumothorax (such as severe COPD (Chronic Obstructive Pulmonary Disease) or extensive emphysema)
* Untreated pneumothorax
* Symptomatic airway obstruction

Discontinuation criteria during ongoing study intervention:

* Heart rate > 120 beats/min
* Systolic blood pressure > 180 mmHg
* Inspired oxygen fraction > 70%
* Respiratory rate > 35/min
* RASS (Richmond Agitation Sedation Scale) ≥ 2
* Doubling of norepinephrine dose or increase of norepinephrine dose to > 0.5 µg/kg/min to maintain mean arterial pressure
* Bradycardia < 45 beats/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Inspiratory effort | Measured during 5 uninterrupted breaths 10 minutes after application of interventional PEEP level
  Inspiratory effort will be measured by the tidal change in esophageal pressure (in cmH2O) during assisted breathing. The esophageal pressure will be measured using a high-resolution manometry catheter. The change from expiratory to inspiratory esophageal pressure will represent the tidal change and be used to estimate the inspiratory effort.
Inspiratory drive | Measured during 5 uninterrupted breaths 10 minutes after application of interventional PEEP level
  The electric activity of the diaphragm (Eadi) will be measured using a NAVA (neurally adjusted ventilatory assist) catheter. The change from end-expiratory to inspiratory Eadi will be calculated. This represents the inspiratory drive. The Eadi will be measured in Voltage.
Effort-to-drive ratio | Calculated from the measures collected 10 minutes after application of interventional PEEP level
  The effort-to-drive ratio (EDR) will be calculated as the inspiratory effort (tidal change in esophageal pressure) divided by the inspiratory drive (tidal change in electric activity of the diaphragm).
Neuromechanical efficiency | Calculated from the measures collected during the occlusion manoeuvre performed 10-15 minutes after application of interventional PEEP level
  The neuromechanical efficiency will be calculated as the change in airway pressure during an occlusion test (Pocc) (measured from end-expiration to maximum negative pressure during the occlusion manoeuvre) divided by the inspiratory change in electric activity of the diaphragm (from end-expiration to inspiration).
Thickening fraction of the diaphragm (TFdi) | Measured 10 minutes after application of interventional PEEP level
  Measured by ultrasound at the right hemidiaphragm. The thickening fraction of the diaphragm (TFdi) will be calculated as [ (end-inspiratory diaphragm thickness - end-expiratory diaphragm thickness) / end-expiratory diaphragm thickness) ].
Transpulmonary driving pressure | Measured during 5 breaths 10 minutes after application of interventional PEEP level
  Change in transpulmonary pressure ( airway pressure - esophageal pressure) from end-expiration to end-inspiration will be calculated using ventilator data and high-resolution manometry
Occlusion pressure | The occlusion pressure will be measured during an occlusion manoeuvre performed 10-15 minutes after application of interventional PEEP level.
  The airway pressure drop from end-expiration to minimum pressure during an occlusion manoeuvre will be measured using the ventilator. The pressure drop indicates the inspiratory effort. It will be measured in cmH2O.

SECONDARY OUTCOMES:
Airway driving pressure | Measured during an inspiratory hold performed 10-15 minutes after application of interventional PEEP level
  Difference in airway pressure between end-expiration and during an inspiratory hold will be calculated from the ventilator data.
Lung compliance | Measured during an inspiratory hold performed 10 - 15 minutes after application of interventional PEEP level
  Lung compliance will be calculated as the tidal volume divided by the change in transpulmonary pressure from end-expiration to end-inspiration.
Thickening fraction of the expiratory abdominal muscles (TFabd) | Measured 10 minutes after application of interventional PEEP level
  The abdominal muscles will be visualized by ultrasound in the anterior axillary line, midway between the inferior border of the ribcage and the iliac crest. The thickening fraction will be calculated as [(expiratory thickness - end-inspiratory thickness) / end-inspiratory thickness ].
Oxygenation | The blood gas will be collected 10 minutes after application of interventional PEEP level
  The PFI (PaO2/FiO2 ratio) will be calculated as arterial PaO2 (partial pressure of oxygen) divided by the FiO2 (fraction of inspired oxygen)
Respiratory system compliance | Measured during an inspiratory hold manoeuvre performed 10-15 minutes after the application of interventional PEEP level.
  The respiratory system compliance will be calculated as the tidal volume divided by the airway driving pressure during an inspiratory hold.

OTHER OUTCOMES:
Central venous oxygen saturation (ScvO2) | Venous blood gas will be collected 10 minutes after application of interventional PEEP level
  Oxygen saturation of venous blood drawn from a central venous catheter.
Tidal volume | Measured in 5 breaths 10 minutes after the application of interventional PEEP level.
  The volume change from end-expiration to end-inspiration. Will be acquired from the ventilator.
Respiratory rate | Measured 10 minutes after the application of interventional PEEP level.
  The number of breaths per minutes (respiratory rate) will be calculated from the volume-time curve acquired from the ventilator.
Dead space | The dead space will be calculated 10 minuted after application of interventional PEEP level.
  Dead space (volume of gas not participating in gas exchange) will be calculated from the difference between arterial and end-expiratory partial pressure of Carbon dioxide, using blood gas analysis and capnography.
Change in end-expiratory lung volume | Measured in the 15 breaths following a PEEP change.
  The change in end-expiratory lung volume will be calculated as the accumulated difference in inspired and expired gas volume during the first 15 breaths after a PEEP change. This will be acquired using the ventilator.
End-expiratory diaphragm thickness | This will be measured during end-expiration 10 minutes after the application of interventional PEEP level.
  The end-expiratory diaphragm thickness will be measured by ultrasound as the thickness of the diaphragm at the right hemisphere at end-expiration.
Neuroventilatory efficiency | Measured from 5 breaths 10 minutes after the application of interventional PEEP level.
  The neuroventilatory efficiency will be calculated as the tidal volume divided by the change from end-expiratory to inspiratory electric activity of the diaphragm (Eadi). The tidal volume will be calculated using data from the ventilator and Eadi acquired using a NAVA (neurally adjusted ventilatory assist) catheter.
Neuromuscular efficiency | This will be calculated from 5 breaths acquired 10 minutes after the application of interventional PEEP level.
  The neuromuscular efficiency will be calculated as the change in transdiaphragmatic pressure (esophageal pressure - gastric pressure) from end-expiration to inspiration divided by the change in electric activity of the diaphragm from end-expiration to inspiration.
Electric activity of the diaphragm | Measured during 5 breaths 10 minutes after application of interventional PEEP level. Additionally measured during an occlusion manoeuvre 10-15 minutes after application of interventional PEEP level.
  Electric activity of the diaphragm (Eadi) during end-expiration, inspiration and occlusion manoeuvres will be measured by NAVA (neurally adjusted ventilator assist) catheters in Voltages
Thickening fraction of the intercostal muscles | Measured 10 minutes after application of interventional PEEP level
  Intercostal muscles will be examined by ultrasound in the cranio-caudal direction at the second intercostal space. The thickening fraction of the intercostal muscles (TFic) will be calculated as the [ (end-inspiratory intercostal thickness - end-expiratory intercostal thickness) / end-expiratory intercostal thickness) ].

CONTACTS AND LOCATIONS:
Overall Officials: Hannes Widing, Principal Investigator — Anesthesia and intensive care medicine, Område 5, Sahlgrenska University hospital, Västra Götalandsregionen
Locations (2):
- Sweden (2):
  - Central intensivvårdsavdelning, Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - Thorax intensivvårdsavdelning, Område 6, Sahlgrenska University Hospital, Västra Götalandsregionen, Gothenburg, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No
The acquired swedish ethical permit does not allow for the sharing of data to international researcher without a confidentiality review or the application of a new ethical permit